CLINICAL TRIAL: NCT05963958
Title: HD-Tdcs Associated With The Use Of Dexmedetomidine For Delirium In Critical Patients With Covid-19
Brief Title: HD-Tdcs and Pharmacological Intervention For Delirium In Critical Patients With COVID-19
Acronym: COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suellen Andrade (Other)
Collaborators: City University of New York (Other)
Responsible Party: Sponsor-Investigator, Suellen Andrade, Principal Investigator, Federal University of Paraíba
Organization: Federal University of Paraíba (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Delirium/HD-tDCS
Record Dates: First submitted 2023-07-01; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: COVID-19; Delirium; Critical Illness
MeSH Terms: conditions — COVID-19; Delirium; Critical Illness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Applicators were blinded to who was receiving active stimulation and who was receiving placebo. The study drug was prepared by the nurses or nursing technicians, or an otherwise uninvolved research associate so that investigators and clinicians were fully masked to allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active HD-tDCS (Experimental): HD-tDCS is delivered on 10 consecutive weekdays, with two sessions per day (in the morning and in the afternoon). For each participant, a 3-mA current is applied via a center anode. The electric current was supplied to the active group and presented an acceleration time of 30 s, maintained at 3 mA for 30 min and then reduced for 30 s. And a maintenance dosage of dexmedetomidine (0.2 - 0.7 mcg/kg per hour).
  Interventions: Combination Product: Active HD-tDCS
- Sham HD-tDCS (Placebo Comparator): HD-tDCS is delivered on 10 consecutive weekdays, with two sessions per day (in the morning and in the afternoon). For the simulated condition, the investigators maintained the same 30-second acceleration up to a total of 3 mA, followed immediately by a 30-second deceleration. And a maintenance dosage of dexmedetomidine (0.2 - 0.7 mcg/kg per hour).
  Interventions: Combination Product: Sham HD-tDCS

INTERVENTIONS:
Combination Product: Active HD-tDCS — Brain stimulation using active high definition transcranial direct current stimulation is applied simultaneously with the use of dexmedetomidine as a pharmacological treatment for delirium in critical illness patients with covid-19
  Arms: Active HD-tDCS
Combination Product: Sham HD-tDCS — Sham high definition transcranial direct current stimulation is applied simultaneously with the use of dexmedetomidine as a pharmacological treatment for delirium in critical illness patients with covid-19
  Arms: Sham HD-tDCS

SUMMARY:
The goal of this clinical trial Is conducted to evaluate the efficacy and safety of active or sham HD-tDCS in combination with dexmedetomidine in patients with moderate to severe ARDS due to COVID-19 with delirium in intensive care unit (ICU). The hypothesis was that HD-tDCS combined with concomitant dexmedetomidine would reduce delirium rates.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years,
* confirmed clinical diagnosis for SARS-CoV-2,
* delirium confirmed through the CAM-ICU-7 test, applied by trained evaluators

Exclusion Criteria:

* severe psychiatric illness that is not well controlled;
* pregnancy or active lactation,
* refusal of consent
* contraindications for brain stimulation such as: aneurysm clips, pacemaker, epilepsy, dermatitis at the site of stimulation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Delirium Severity | 28 days
  delirium severity over the 28-day study period is measured using the CAM-ICU-7. Patients discharged before 28 days were considered without delirium.

SECONDARY OUTCOMES:
length of stay in the ICU and hospital stay | 28 days
  defined as the total number of days that patients remained in the hospital from the date of randomization to the date of hospital discharge
Occurrence of hypotension requiring any vasopressor administration | 28 days
C-reactive protein levels | 28 days
ventilator-free days during the first 28 days | 28 days
  defined as the number of days free from mechanical ventilation for at least 48 consecutive hours
Exploratory analisys | 28 days
  Organ dysfunction and clinical response; use of Concomitant Medications; Richmond Agitation Sedation Scale (RASS) and mortality prognosis

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Paraiba, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: No